CLINICAL TRIAL: NCT01548183
Title: Mobile Phone Text-message Program to Reduce Risky Sexual Behavior in Young Females Discharged From the Emergency Department
Brief Title: Text-message Program to Reduce Risky Sexual Behavior in Young Adult Female Emergency Department (ED) Patients
Acronym: StARSS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PRO10100400
Record Dates: First submitted 2012-02-22; First posted 2012-03-08 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Education, Sex
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle counseling (Experimental): Weekly SMS assessing risky sexual encounters and providing feedback including concern, goal-setting and tools to reduce risk
  Interventions: Behavioral: Lifestyle counseling
- Usual care (No Intervention): Usual care includes ED provider counseling as per normal clinical care

INTERVENTIONS:
Behavioral: Lifestyle counseling — Weekly SMS assessments of risky sexual encounters with feedback
  Arms: Lifestyle counseling

SUMMARY:
The US preventative services task force (USPSTF) recommends behavioral counseling in the primary care setting for prevention of sexually transmitted diseases, however, screening and counseling rarely occur. Text messaging (TM) is increasingly being used as a tool to affect behavior change in patients, but its effect on patients that report at-risk sexual behavior in the emergency department (ED) is unknown. The investigators seek to assess the feasibility of ED-based screening of young adult females for at-risk sexual behavior and enrolling them in a 3 month trial using TM to deliver information and skill building to improve health behavior.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18-25 years
* AUDIT-C score > 2
* (Drugs or alcohol prior to last sex OR No condom with last sex OR > 1 partner in last 3 months)

Exclusion Criteria:

* No personal cell phone with SMS features
* Prisoner
* Pregnant or planning in next 3 months
* Current or past drug/alcohol treatment or psychiatric treatment

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2011-08; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Sex without condom | 3 months after ED discharge
  Participants will be called for phone follow-up at 12 weeks post-ED discarge

SECONDARY OUTCOMES:
Number of unprotected vaginal sexual encounters | 3 months post-ED discharge
  Participants will be called for phone follow-up at 12 weeks post ED discharge

CONTACTS AND LOCATIONS:
Locations (1):
- UPMC Mercy Hospital, Pittsburgh, Pennsylvania, United States